CLINICAL TRIAL: NCT02213900
Title: Preventing Post-Operative Delirium in Pneumonectomy, Esophagectomy and Thoracotomy Patients
Brief Title: Preventing Post-Operative Delirium in Patients Undergoing a Pneumonectomy, Esophagectomy or Thoracotomy
Acronym: PE-POD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Principle Investigator, Regenstrief Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VFR-398-Khan
Record Dates: First submitted 2014-03-18; First posted 2014-08-12 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Delirium; Cognitive Impairment; Post-traumatic Stress Disorder; Depression; Anxiety
Keywords: delirium; confusion; surgery; cognitive Impairment; post-traumatic Stress disorder; depression; anxiety
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Confusion | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haloperidol (Experimental): Randomized patients will receive 0.5mg Haloperidol immediately after surgery and Q8H following the initial dose for a total of 4 days.
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator): Randomized patients will receive a placebo solution immediately after surgery and Q8H following for a total of 4 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — 0.5mg IV Push immediately after surgery and Q8H following for a total of 4 days
  Arms: Haloperidol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effectiveness of a preventative low-dose of Haloperidol to prevent delirium in patients undergoing a esophagectomy, pneumonectomy or thoracotomy.

Delirium is state of severe confusion and some symptoms include:

* Cannot think clearly
* Have trouble paying attention
* Have a hard time understanding what is going on around them
* May see or hear things that are not there. These things seem very real to them.

DETAILED DESCRIPTION:
50% of patients who undergo esophageal and/or lung resection suffer from acute brain dysfunction or delirium postoperatively. Delirium is a state of brain failure characterized by disturbance of consciousness with reduced ability to focus, sustain, or shift attention that occurs over a short period of time and tends to fluctuate over the course of the day. Presence of delirium in the post-operative phase is associated with a longer length of both intensive care unit and hospital stay, increased health-care costs, long-term functional and cognitive decline, and an increased risk of in-hospital and post-discharge mortality.

Haloperidol primarily acts by blocking dopamine (D2) receptors. This dopamine blockade in the cerebral cortex improves cognition and reduces delirium. Along with the dopamine blockade, haloperidol has anti-inflammatory properties. It inhibits production of lipopolysaccharide induced pro-inflammatory cytokines, interleukin (IL-1) and tumor necrosis factor alpha (TNF-α). Haloperidol also increases levels of Interleukin -1 receptor antagonist (IL-1RA), an anti-inflammatory cytokine that blocks the action of other pro-inflammatory cytokines. If unchecked, the inflammatory cytokines cause impaired concentration, sleep disturbances, and agitation the cardinal symptoms of delirium; and induce a reduction in cholinergic activity. Given the inhibitory effect of acetylcholine on certain cytokines such as interleukin-6, a repetitive cycle of inadequate regulation of inflammation due to cholinergic depletion ensues. Haloperidol with its anti-inflammatory properties seeks to mitigate this repetitive vicious cycle.

ELIGIBILITY:
Inclusion Criteria:

1. At least ≥ 18 years of age and older
2. Undergoing a possible or scheduled thoracotomy
3. English speaking

Exclusion Criteria:

1. History of Schizophrenia and Parkinson's disease
2. History of Severe Dementia
3. History of Alcohol Abuse
4. On Cholinesterase Inhibitors or Levodopa
5. Pregnant or Nursing
6. Corrected QT interval > 550 milliseconds at the time of randomization
7. History of Neuroleptic Malignant Syndrome or Haloperidol Allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babar A Khan, MD, MS, Principal Investigator — Regenstrief Institute, Inc.; Kenneth A Kesler, MD, Principal Investigator — IU School of Medicine
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Khan BA, Perkins AJ, Campbell NL, Gao S, Khan SH, Wang S, Fuchita M, Weber DJ, Zarzaur BL, Boustani MA, Kesler K. Preventing Postoperative Delirium After Major Noncardiac Thoracic Surgery-A Randomized Clinical Trial. J Am Geriatr Soc. 2018 Dec;66(12):2289-2297. doi: 10.1111/jgs.15640. Epub 2018 Nov 21. PMID 30460981

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Randomized patients will receive a placebo solution immediately after surgery and Q8H following for a total of 4 days.
  Placebo
Period: Overall Study
Arm/Group | Haloperidol | Placebo
Started | 68 | 67
Completed | 68 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol | Placebo | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (12.4) | 59.6 (14.0) | 59.6 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 46 | 54 | 100

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Low-dose Haloperidol in Reducing Delirium Incidence
Description: Test the efficacy of low dose haloperidol in reducing delirium incidence among patients who are status post esophagectomy, pneumonectomy or thoracotomy compared to placebo.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol | Placebo
Number analyzed (Participants) | 68 | 67
Participants | 15 | 19

2. Secondary Outcome: Efficacy of Low-dose Haloperidol in Reducing Days With Delirium
Description: Test the efficacy of low dose haloperidol in reducing the number of days with delirium among patients who are status post esophagectomy, pneumonectomy or thoracotomy compared to placebo.
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Days with Delirium
Arm/Group | Haloperidol | Placebo
Number analyzed (Participants) | 68 | 67
Days with Delirium | 0.3 (0.7) | 0.5 (0.9)

3. Secondary Outcome: Efficacy of Low-dose Haloperidol in Reducing ICU and Hospital Length of Stay
Description: Test the efficacy of low dose haloperidol in reducing ICU and hospital length of stay among patients who are status post esophagectomy or pneumonectomy compared to placebo.
Time Frame: Date of hospital admission through date of hospital discharge, up to 3 weeks on average.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Haloperidol | Placebo
Number analyzed (Participants) | 68 | 67
Days
  ICU Length of Stay | 2.5 (2.2) | 2.8 (10.2)
  Overall Length of Stay | 9.3 (3.5) | 10.2 (4.6)

4. Secondary Outcome: Efficacy of Low-dose Haloperidol in Reducing Cognitive Impairment at Post-operative Follow-up
Description: Test the efficacy of low dose haloperidol in reducing cognitive impairment at post-operative follow-up among patients who are status post esophagectomy, pneumonectomy or thoracotomy compared to placebo. Cognitive status is assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The RBANS measures attention, language, visuospatial/constructional abilities, and memory. It is made up of 12 subtests. The subtests produce 5 index scores and a total scale score. All the subtest scores are summed to calculate a Total Index score. The Total Index score is presented. The Total Index score scale is from 0-100 with higher scores indicating less cognitive impairment.
Time Frame: Up to 3 months after hospital discharge on average.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Haloperidol | Placebo
Number analyzed (Participants) | 68 | 67
Units on a scale
  Baseline RBANS Total Score | 31.7 (27.6) | 30.1 (22.8)
  3 Month RBANS Total Score | 31.8 (30.1) | 22.7 (23.2)

ADVERSE EVENTS:
Arm/Group | Haloperidol | Placebo
Serious Adverse Events (participants affected / at risk) | 3/68 | 2/67
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haloperidol (N=68) | Placebo (N=67)
Death (General disorders) | 0 (0) | 1 (1)
Life Threatening Episode (General disorders) | 1 (1) | 1 (1)
Inpatient or Prolonged Current Hospitalization (General disorders) | 2 (2) | 0 (0) — Could include significant incapacitation or an episode requiring intervention to prevent permanent impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No